CLINICAL TRIAL: NCT03798080
Title: A Randomized, 30-week, Active-controlled, Open-label, 2 Treatment-arm, Parallel Group, Multicenter Study Comparing Efficacy and Safety of iGlarLixi to Insulin Glargine With or Without Metformin in Patients With Type 2 Diabetes Mellitus Insufficiently Controlled on Basal Insulin With or Without Oral Antidiabetic Drug(s)
Brief Title: Comparison of the Efficacy and Safety of Insulin Glargine/Lixisenatide Fixed Ratio Combination to Insulin Glargine in Patients With Type 2 Diabetes Insufficiently Controlled on Basal Insulin
Acronym: Lixilan-L-CN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14944; U1111-1190-7781 (Other: UTN)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Soliqua (insulin glargine/lixisenatide) (Experimental): iGlarLixi (insulin glargine/lixisenatide) will be self-administered subcutaneously once daily in the morning with or without metformin for 30 weeks
  Interventions: Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010); Drug: Metformin
- Lantus (insulin glargine) (Active Comparator): Insulin glargine will be self-administered subcutaneously once daily at any time of the day with or without metformin for 30 weeks
  Interventions: Drug: Insulin glargine (HOE901); Drug: Metformin

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Soliqua; iGlarLixi
  Arms: Soliqua (insulin glargine/lixisenatide)
Drug: Insulin glargine (HOE901) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Lantus (insulin glargine)
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To demonstrate the superiority of iGlarLixi (fixed ratio combination of insulin glargine and lixisenatide) to insulin glargine on glycemic control as assessed by glycated hemoglobin A1c (HbA1c) change in patients with type 2 diabetes mellitus (T2DM) who are not sufficiently controlled with basal insulin.

Secondary Objectives:

* To assess the effects of iGlarLixi in comparison with insulin glargine
* To assess the safety in each treatment group

DETAILED DESCRIPTION:
The maximum study duration per patient will be approximately 33 weeks: an up to 2-week screening period (it can be exceptionally extended up to one additional week), a 30-week, open label randomized treatment period comparing iGlarLixi to insulin glargine (± metformin for both treatments), and a 3-day post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year and treated with basal insulin for at least 6 months before screening visit (V1).
* Patients who have been treated with a stable basal insulin regimen (ie, type of insulin and time/frequency of the injection), for at least 3 months before screening visit (V1).
* Stable total daily basal insulin dose (±20 %) in the range of 10 and 25 U/day for at least 2 months before screening visit (V1). Total daily dose should be within the range of 10-25 U, both inclusive, on the day of screening, but individual fluctuations of ±20% within 2 months prior to screening are acceptable.
* For patients receiving basal insulin AND 1 or 2 oral anti-diabetic drugs (OADs): the OAD dose(s) must be stable during the 3 months prior to screening. The OAD(s) can be 1 to 2 out of:
* Metformin (≥1500 mg/day or maximal tolerated dose).
* Sulfonylurea (SU)/glinide.
* Alpha-glucosidase inhibitor (alpha-GI).
* Sodium-glucose co-transporter 2 (SGLT2) inhibitor.
* Dipeptidyl-peptidase-4 (DPP-4) inhibitor.
* Fasting plasma glucose (FPG) ≤160 mg/dL (8.9 mmol/L) at screening visit (V1) (can be repeated once to confirm).
* Signed written informed consent.

Exclusion criteria:

* Age <18 years at screening visit (V1).
* Screening glycated hemoglobin A1c(HbA1c) <7.0% or >10.5%.
* History of hypoglycemia unawareness.
* History of metabolic acidosis, including diabetic ketoacidosis within one year prior to screening.
* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria within 3 months prior to screening.
* Previous use of insulin regimen other than basal insulin, eg, prandial or pre-mixed insulin, within one year prior to screening (Note: Short term treatment [≤10 days] due to intercurrent illness is allowed).
* History of discontinuation of a previous treatment with glucagon-like-peptide-1 receptor agonists (GLP-1 RAs) due to safety/tolerability reason or lack of efficacy.
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to screening.
* Use of weight loss drugs within 3 months prior to screening.
* Use of any investigational drug within 1 month or 5 half-lives, whichever is longer, prior to screening.
* Within 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization.
* Planned coronary, carotid, or peripheral revascularization procedures to be performed during the study period.
* Known history of drug or alcohol abuse within 6 months prior to screening.
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure >180 mmHg or diastolic blood pressure >95 mmHg.
* Laboratory findings at screening visit:
* Amylase and/or lipase >3 times the upper limit of normal (ULN) laboratory range.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN.
* Total bilirubin >1.5 ULN (except in case of Gilbert's syndrome).
* Calcitonin ≥20 pg/mL (5.9 pmol/L).
* Hemoglobin <10.5 g/dL and/or neutrophils <1500/mm3 and/or platelets <100 000/mm3.
* Positive test for hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody (HCAb).
* Positive urine pregnancy test in female of childbearing potential.
* For patient not treated with metformin at screening: severe renal function impairment with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 or end-stage renal disease.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (ie, worsening) or not controlled (ie, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening visit; or history of surgery affecting gastric emptying.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes).
* Mean fasting self-monitored plasma glucose (SMPG) is >160 mg/dL (8.9 mmol/L), calculated from all available (minimum of 4 self-measurements) values during the 7 days prior to randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From Baseline to Week 30
  Change in glycated hemoglobin (HbA1c) from baseline to Week 30

SECONDARY OUTCOMES:
Patients with HbA1c <7.0% | At Week 30
  Percentage of patients reaching HbA1c <7% at Week 30
Patients with HbA1c ≤ 6.5% | At Week 30
  Percentage of patients reaching HbA1c ≤ 6.5% at Week 30
Change in postprandial plasma glucose (PPG) | From Baseline to Week 30
  Absolute change in 2-hour blood glucose excursion and PPG during meal test from baseline to Week 30
Change in self-monitored plasma glucose (SMPG) profile | From Baseline to Week 30
  Absolute change in 7-point SMPG profiles from baseline to Week 30 (each time point and average daily value)
Patients with HbA1c <7.0% with no body weight gain | At Week 30
  Percentage of patients reaching HbA1c <7% with no body weight gain at Week 30
Change in body weight | From Baseline to Week 30
  Absolute change in body weight from baseline to Week 30
Patients with HbA1c <7.0% with no body weight gain and no documented symptomatic hypoglycemia | At Week 30
  Percentage of patients reaching HbA1c <7% with no body weight gain at Week 30 and no documented (plasma glucose [PG] ≤70 mg/dL [3.9mmol/L]) symptomatic hypoglycemia during the 30-week randomized treatment period
Patients requiring rescue therapy | From Baseline to Week 30
  Percentage of patients requiring rescue therapy during the 30-week randomized treatment period
Change in fasting plasma glucose (FPG) | From Baseline to Week 30
  Absolute change in FPG from baseline to Week 30
Confirmed hypoglycemia | From Baseline to Week 30
  Severe hypoglycemia and episodes of hypoglycemia documented with PG ≤ 70 mg/dL (3.9mmol/L) regardless of symptoms
Adverse events (AEs) | From Baseline to Week 30
  Number of AEs, Serious AEs, AEs of Special Interest, and AEs requiring specific monitoring from baseline to Week 30
Immunogenicity (antibody variables) | From Baseline to Week 30
  Anti-lixisenatide antibodies (in iGlarLixi group) and anti-insulin antibodies from baseline to Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (45):
- China (45):
  - Investigational Site Number 1560044, Baotou
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560039, Beijing
  - Investigational Site Number 1560005, Changchun
  - Investigational Site Number 1560054, Changchun
  - Investigational Site Number 1560015, Changsha
  - Investigational Site Number 1560010, Chenzhou
  - Investigational Site Number 1560030, Chongqing
  - Investigational Site Number 1560025, Fuzhou
  - Investigational Site Number 1560016, Guangzhou
  - Investigational Site Number 1560053, Guangzhou
  - Investigational Site Number 1560045, Guangzhou
  - Investigational Site Number 1560021, Hefei
  - Investigational Site Number 1560018, Hohhot
  - Investigational Site Number 1560019, Huanggang
  - Investigational Site Number 1560041, Jiaxing
  - Investigational Site Number 1560040, Jinan
  - Investigational Site Number 1560007, Jinan
  - Investigational Site Number 1560026, Jinzhou
  - Investigational Site Number 1560042, Kaifeng
  - Investigational Site Number 1560003, Kunming
  - Investigational Site Number 1560032, Lanzhou
  - Investigational Site Number 1560033, Luoyang
  - Investigational Site Number 1560028, Nanjing
  - Investigational Site Number 1560013, Nanjing
  - Investigational Site Number 1560017, Nanjing
  - Investigational Site Number 1560035, Nanjing
  - Investigational Site Number 1560038, Nanjing
  - Investigational Site Number 1560046, Nantong
  - Investigational Site Number 1560008, Pingxiang
  - Investigational Site Number 1560037, Qingdao
  - Investigational Site Number 1560031, Qinhuangdao
  - Investigational Site Number 1560011, Shanghai
  - Investigational Site Number 1560002, Shanghai
  - Investigational Site Number 1560027, Shanghai
  - Investigational Site Number 1560047, Shanghai
  - Investigational Site Number 1560012, Shenyang
  - Investigational Site Number 1560006, Tianjin
  - Investigational Site Number 1560049, Ürümqi
  - Investigational Site Number 1560020, Xining
  - Investigational Site Number 1560050, Xining
  - Investigational Site Number 1560036, Xuzhou
  - Investigational Site Number 1560023, Yangzhou
  - Investigational Site Number 1560022, Zhuzhou
  - Investigational Site Number 1560052, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Yuan X, Guo X, Zhang J, Dong X, Lu Y, Pang W, Gu S, Niemoeller E, Ping L, Nian G, Souhami E; LixiLan-L-CN investigators. Improved glycaemic control and weight benefit with iGlarLixi versus insulin glargine 100 U/mL in Chinese people with type 2 diabetes advancing their therapy from basal insulin plus oral antihyperglycaemic drugs: Results from the LixiLan-L-CN randomized controlled trial. Diabetes Obes Metab. 2022 Nov;24(11):2182-2191. doi: 10.1111/dom.14803. Epub 2022 Jul 25. PMID 35762489
- [Derived] Yuan X, Li D, Wang K, Lauand F, Zhang M, Fang H, Du Q, Kang L, Alvarez A, Guo X. iGlarLixi effectively reduces residual hyperglycaemia in Chinese people with type 2 diabetes on basal insulin: A post hoc analysis of the LixiLan-L-CN study. Diabetes Obes Metab. 2024 Dec;26(12):5942-5949. doi: 10.1111/dom.15968. Epub 2024 Oct 3. PMID 39360440
- [Derived] Guo X, Yang W, Zhang J, Dong X, Liu M, Gu S, Lauand F, Li L, Huang Q, Kang L, Souhami E. iGlarLixi provides a higher derived time-in-range versus insulin glargine 100 U/mL or lixisenatide in Asian Pacific people with type 2 diabetes: A post hoc analysis. Diabetes Obes Metab. 2023 Jul;25(7):2005-2011. doi: 10.1111/dom.15074. Epub 2023 May 3. PMID 36999231